CLINICAL TRIAL: NCT03893565
Title: A Multicentre Randomized, Double-blind, Placebo-controlled Phase 2 Study to Evaluate the Safety, Tolerability, Efficacy, Dose-response, Pharmacokinetics and Pharmacodynamics of Repeat Dosing of an Anti-LAG3 Cell Depleting Monoclonal Antibody (GSK2831781) in Patients With Active Ulcerative Colitis
Brief Title: Safety, Tolerability, Efficacy and Dose-response of GSK2831781 in Ulcerative Colitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was stopped based on the assessment of clinical data.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 204869
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Results first posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-03

CONDITIONS: Colitis, Ulcerative
Keywords: GSK2831781; Ulcerative colitis; Anti-LAG3 cell Depleting monoclonal antibody; Dose-response
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: This is a parallel group, placebo controlled study where participants will be randomized to receive either GSK2831781 or placebo.
Who Masked: Participant, Investigator
Masking Description: This will be a double-blind study. Induction doses will be matched with placebo. For Maintenance dosing, participant and investigator will be masked. Participants will be allocated to the next treatment phase according to their Responder status. Non-responders to the double-blind Induction Phase will receive treatment in Open-Label Induction phase where there will be no masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- GSK2831781-Double blind phase (Experimental): Eligible participants will receive GSK2831781 intravenously in the double blind induction phase at different dose levels. Participants identified as Responders at Week 10 will then receive GSK2831781 subcutaneously during the double-blind ETP from Week 14 until Week 26
  Interventions: Drug: GSK2831781 - Double Blind Phase
- GSK2831781- Open label phase (Experimental): Eligible participants will receive GSK2831781 intravenously in the open label induction phase. Participants identified as Non-Responders at Week 10 will receive GSK2831781 from Week 12 until Week 22. Participants identified as Responders at Week 22 will enter open label ETP to receive GSK2831781 from Week 26 until Week 38. Participants identified as Non- Responders at Week 22 will discontinue treatment.
  Interventions: Drug: GSK2831781 - Open Label phase
- Placebo matching GSK2831781- Double blind phase (Placebo Comparator): Eligible participants will receive Placebo in the double blind induction phase Participants identified as Responders at Week 10 will continue to receive Placebo subcutaneously during the double-blind ETP from Week 14 until Week 26.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK2831781 - Double Blind Phase — GSK2831781 will be administered intravenously in the double blind induction phase and subcutaneously in the double blind ETP (both according to randomization).
  Arms: GSK2831781-Double blind phase
Drug: Placebo — Placebo (commercial saline solution) will be administered intravenously in the double blind induction phase and subcutaneously in the double blind ETP (both according to randomization).
  Arms: Placebo matching GSK2831781- Double blind phase
Drug: GSK2831781 - Open Label phase — GSK2831781 will be administered intravenously in the open label induction phase and subcutaneously in the open label ETP.
  Arms: GSK2831781- Open label phase

SUMMARY:
This is a Phase 2, multicenter, randomized, double-blind, parallel group, placebo-controlled study to investigate the safety, tolerability, efficacy and dose-response of GSK2831781 in participants with moderate to severe active ulcerative colitis. The study consists of a 5-week screening window, 10-week Induction Phase, 30-week double-blind Extended Treatment Phase (ETP) with 42-week Follow-Up Phase. Non-Responders identified following the Week 10 assessment will be allocated to open label treatment, consisting of Induction (Weeks 12 to 22), an Open label ETP (Weeks 22 to 42) and a follow-Up to Week 54.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years of age or older and > 40 kilograms (kg) at the time of signing the informed consent.
* Participants who have a diagnosis of ulcerative colitis, established at least 3 months prior to screening, as documented by diagnostic sigmoidoscopy or colonoscopy, and biopsy.
* Complete 4-domain Mayo Score of 6 to 12, with disease extending >= 15 centimeters (cm) from the anal verge, with a centrally read endoscopic sub score of >=2 at screening endoscopy, and a rectal bleeding sub score >=1.
* A history of at least one of the following: inadequate response to, loss of response to, or intolerance to azathioprine or mercaptopurine (including thiopurine methyltransferase [TPMT] and nudix hydrolase 15 [NUDT15] genetic mutations precluding use), ciclosporin, tacrolimus or methotrexate; inadequate response to, loss of response to, intolerance to, or demonstrated dependence on oral corticosteroids; inadequate response to, loss of response to, or intolerance to at least one approved advanced therapy for UC including anti- tumor necrosis factor (TNF) therapies (example given [e.g.] infliximab, adalimumab, golimumab, or biosimilar), anti-integrin therapies, anti-interleukin (IL)-12/23 monoclonal antibodies or Janus Kinase (JAK) inhibitors.
* Surveillance colonoscopy (performed according to local standards) within 12 months of screening (or during screening, if required) for participants with: Pancolitis of >8 years duration; or participants with left-sided colitis of >12 years duration. For participants for whom this criterion does not apply, colorectal cancer surveillance should be undertaken according to local or national guidelines for participants with age >=50, or with other known risk factors for colorectal cancer.
* Both male and female participants are eligible to participate.
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: Not a woman of childbearing potential (WOCBP); A WOCBP who agrees to use a highly effective contraceptive method for at least 4 weeks prior to dosing, until the Follow-Up visit.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Participants with a current diagnosis of indeterminate colitis, inflammatory bowel disease-unclassified, Crohn's disease, infectious colitis, or ischemic colitis.
* Participants with fulminant ulcerative colitis (as defined by 6 bloody stools daily and 1 or more of body temperature >=100.4 degrees Fahrenheit (or 38 degree Celsius) or heart rate >90 beats per minute), or toxic megacolon.
* Prior extensive colonic resection, subtotal or total colectomy, or proctocolectomy, or planned surgery for ulcerative colitis.
* Participants with any uncontrolled medical conditions, other than active ulcerative colitis, that in the opinion of the investigator put the participant at unacceptable risk or interfere with study assessments or integrity of the data. Other medical conditions should be stable at the time of screening and be expected to remain stable for the duration of the study.
* Unstable lifestyle factors, such as alcohol use to excess or recreational drug use, to the extent that in the opinion of the investigator they would interfere with the ability of a participant to complete the study.
* An active infection or a history of serious infections as follows: a) Use of antimicrobials (antibacterials, antivirals, antifungals or antiparasitic agents) for an infection within 30 days before first dose (topical treatments may be allowed at the Medical Monitor's discretion). b) A history of opportunistic infections within 1 year of screening (e.g. Pneumocystis jirovecii, aspergillosis or Cytomegalovirus colitis). This does not include infections that may occur in immunocompetent individuals, such as fungal nail infections or vaginal candidiasis, unless it is of an unusual severity or recurrent nature. c) Recurrent or chronic infection or other active infection that, in the opinion of the Investigator, might cause this study to be detrimental to the participant. d) Symptomatic herpes zoster within 3 months prior to screening. e) History of tuberculosis (active or latent), irrespective of treatment status. f) A positive diagnostic tuberculosis test at screening (defined as a positive QuantiFERON test). In cases where the QuantiFERON test is indeterminate, the participant may have the test repeated once and if their second test is negative they will be eligible. In the event a second test is also indeterminate, the investigator has the option to undertake Purified Protein Derivative (PPD) testing. If the PPD reaction is less than (<) 5 millimeter (mm), then the participant is eligible. If the reaction is >= 5mm, or PPD testing is not undertaken, the participant is not eligible. g) Positive Clostridium difficile toxin test during screening. However, rescreening can be undertaken following successful treatment.
* Current or history of chronic liver or biliary disease (with the exception of Gilbert's syndrome, asymptomatic gallstones or uncomplicated fatty liver disease).
* Hereditary or acquired immunodeficiency disorder, including immunoglobulin deficiency (unless the participant has a documented history of selective immunoglobulin A deficiency).
* A major organ transplant (e.g. heart, lung, kidney, liver, pancreas) or hematopoietic stem cell/marrow transplant.
* Any planned major surgical procedure during the study.
* A history of malignant neoplasm within the last 5 years, except for adequately treated non-metastatic basal or squamous cell cancers of the skin (within 1 year) or carcinoma in situ of the uterine cervix (within 3 years) that has been fully treated and shows no evidence of recurrence.
* A change in dose of oral sulfasalazine or aminosalicylate within 2 weeks prior to Baseline endoscopy.
* Greater than 20 mg per day oral prednisolone (or equivalent), or a change in dose of corticosteroid within 2 weeks prior to Baseline endoscopy, or anticipated inability to maintain a stable dose of corticosteroids (<=20 mg oral prednisolone or equivalent) until Week 12.
* Topical (rectal) corticosteroids or topical (rectal) aminosalicylate within 2 weeks prior to Baseline endoscopy.
* Initiation or a change in dose of mercaptopurine or azathioprine (including initiation or discontinuation of allopurinol) or methotrexate within 8 weeks prior to Baseline endoscopy.
* Treatment with ciclosporin, tacrolimus or thalidomide within 4 weeks prior to Baseline endoscopy.
* Treatment with an anti-TNF biologic within 8 weeks prior to Baseline endoscopy, anti-integrin or anti-IL-12/23 biologics within 12 weeks prior to Baseline endoscopy, or a JAK inhibitor within 4 weeks prior to Baseline endoscopy.
* A history of inadequate response, loss of response, or intolerance to more than three classes of approved advanced therapies for UC (including anti-TNF therapies, anti-integrin therapies, anti-IL-12/23 monoclonal antibodies, or JAK inhibitors; but excluding exposure within a clinical trial setting), of which participants must not have had inadequate response (primary non-response) to more than two classes.
* Received fecal microbiota transplantation within 4 weeks prior to Baseline endoscopy.
* Received live vaccination within 4 weeks of Day 1 or plan to receive during the study until Follow-Up.
* The participant has participated in a clinical trial and has received an investigational product within the following time period prior to the screening endoscopy day in the current study:

  1. Biologics: 3 months, 5 half-lives, or twice the duration of the biological effect of the investigational product (whichever is longer);
  2. New Chemical Entities (NCEs): 30 days, 5 half-lives, or twice the duration of the biological effect (whichever is longer).
* Absolute neutrophil count <1.5 times 10^9 cells per liter (L) or a hemoglobin <80 grams per liter (g/L) or lymphocyte count <0.8 times 10^9 cells /L.
* Estimated glomerular filtration rate (GFR) by Chronic Kidney Disease Epidemiology Collaboration equation (CKD-EPI) calculation <60 milliliter (mL) per minute per 1.73 m^2 at screening.
* ALT >2 times upper limit of normal (ULN) and bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent) at screening.
* Other clinically significant abnormalities of laboratory assessments, as judged by the investigator and/or GlaxoSmithKline Medical Monitor that could affect the safety of the participant, or the interpretation of the data from the study.
* Presence of hepatitis B surface antigen (HBsAg) or Hepatitis B core antibody (HBcAb), or positive hepatitis C antibody result at screening (Nota bene [NB]-Participants with Hepatitis C antibody due to prior resolved disease can be enrolled only if a confirmatory negative Hepatitis C ribonucleic acid [RNA] test is obtained).
* Positive serology for human immunodeficiency virus (HIV) at screening.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 3 months.
* QTc >450 milliseconds (msec) or QTc >480 msec for participants with bundle branch block at screening and Day 1. The QTc is the QT interval corrected for heart rate according to either Bazett's formula (QTcB), Fridericia's formula (QTcF), or another method, machine or over read.
* Participants with hypersensitivity to GSK2831781 or any excipients in the clinical formulation of GSK2831781.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (57):
- United States (4):
  - GSK Investigational Site, Northridge, California
  - GSK Investigational Site, Rialto, California
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, San Antonio, Texas
- GSK Investigational Site, Sofia, Bulgaria
- Czechia (3):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Slaný
- GSK Investigational Site, Tallinn, Estonia
- France (5):
  - GSK Investigational Site, Grenoble
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Saint-Priest-en-Jarez
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Vandœuvre-lès-Nancy
- India (5):
  - GSK Investigational Site, Jaipur
  - GSK Investigational Site, Ludhiana
  - GSK Investigational Site, Nagpur
  - GSK Investigational Site, Rajkot
  - GSK Investigational Site, Varanasi
- GSK Investigational Site, Osaka, Japan
- GSK Investigational Site, Amsterdam, Netherlands
- Poland (14):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Elblag
  - GSK Investigational Site, Kamieniec Ząbkowicki
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Knurów
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Rzeszów
  - GSK Investigational Site, Sopot
  - GSK Investigational Site, Staszów
  - GSK Investigational Site, Torun
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
  - GSK Investigational Site, Zamość
- Russia (6):
  - GSK Investigational Site, Krasnoyarsk
  - GSK Investigational Site, Nizhny Novgorod
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Samara
  - GSK Investigational Site, Saratov
- GSK Investigational Site, Zrenjanin, Serbia
- GSK Investigational Site, Prešov, Slovakia
- South Africa (4):
  - GSK Investigational Site, Port Elizabeth, Eastern Cape
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Gauteng
  - GSK Investigational Site, Pretoria
- Ukraine (7):
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Lviv
  - GSK Investigational Site, Odesa
  - GSK Investigational Site, Vinnytsia
  - GSK Investigational Site, Zaporizhzhia
  - GSK Investigational Site, Zaporizhzhya
- United Kingdom (3):
  - GSK Investigational Site, Cambridge, Cambridgeshire
  - GSK Investigational Site, Headington, Oxfordshire
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] D'Haens G, Peyrin-Biroulet L, Marks DJB, Lisi E, Liefaard L, Beaton A, Srinivasan N, Bouma G, Prasad N, Cameron R, Kayali Z, Tarzi R, Hanauer S, Sandborn WJ. A randomised, double-blind, placebo-controlled study of the LAG-3-depleting monoclonal antibody GSK2831781 in patients with active ulcerative colitis. Aliment Pharmacol Ther. 2023 Aug;58(3):283-296. doi: 10.1111/apt.17557. Epub 2023 Jun 16. PMID 37323059

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, placebo-controlled study to evaluate the safety, tolerability, efficacy and dose-response of GSK2831781 in participants with ulcerative colitis. The study was conducted across 13 countries.
Pre-assignment Details: A total of 104 participants were enrolled in the study. This study was terminated based on the assessment of clinical data.
Groups:
- Placebo IV: Participants were administered placebo via the intravenous (IV) route on Day 1, Weeks 2, 6 and 10. At Week 10, participants underwent Induction assessment including endoscopy.
- GSK2831781 450 mg IV: Participants were administered GSK2831781 450 milligrams (mg) via the IV route on Day 1, Weeks 2, 6 and 10. At Week 10, participants underwent Induction assessment including endoscopy.
- GSK2831781 300 mg IV: Participants were administered GSK2831781 300 mg via the IV route on Day 1, Weeks 2, 6 and 10. At Week 10, participants underwent Induction assessment including endoscopy.
- GSK2831781 150 mg IV: Participants were administered GSK2831781 150 mg via the IV route on Day 1, Weeks 2, 6 and 10. At Week 10, participants underwent Induction assessment including endoscopy.
- GSK2831781 45 mg IV: Participants were administered GSK2831781 45 mg via the IV route on Day 1, Weeks 2, 6 and 10. At Week 10, participants underwent Induction assessment including endoscopy.
- Placebo SC: Participants from the placebo arm identified as responders based on Week 10 assessments during the Induction Phase received placebo subcutaneously (SC) every 4 weeks from Weeks 14 to 26 during the 20 week double-blind extended treatment phase (ETP). At Week 30, participants underwent an assessment following which they were followed up until Week 42.
- GSK2831781 300 mg SC: Participants from the GSK2831781 arms identified as responders based on Week 10 assessments during the Induction Phase received GSK2831781 300 mg SC every 4 weeks from Weeks 14 to 26 during the 20-week double-blind ETP. At Week 30, participants underwent an assessment following which they were followed up until Week 42.
- Open-label GSK2831781 450 mg IV: Participants identified as non-responders during the double-blind Induction phase at Week 10 were administered GSK2831781 450 mg IV on Weeks 12, 14, 18 and 22 during the open-label (OL) induction phase.
- Open-label GSK2831781 300 mg SC: Participants from the Open-label induction phase who responded at Week 22 entered the 20-week (Week 22 to Week 42) open-label extended treatment phase and received GSK2831781 300 mg SC every 4 weeks from Week 26 until Week 38. Participants were followed up until Week 54.
Period: Double-blind Induction Phase (10 Weeks)
Arm/Group | Placebo IV | GSK2831781 450 mg IV | GSK2831781 300 mg IV | GSK2831781 150 mg IV | GSK2831781 45 mg IV | Placebo SC | GSK2831781 300 mg SC | Open-label GSK2831781 450 mg IV | Open-label GSK2831781 300 mg SC
Started | 27 | 48 | 11 | 10 | 8 | 0 | 0 | 0 | 0
Completed | 21 | 32 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Not Completed | 6 | 16 | 10 | 9 | 7 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 6 | 0 | 0 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 5 | 5 | 9 | 0 | 6 | 0 | 0 | 0 | 0
Not completed — Protocol-specified withdrawal criterion met | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Period: Double-blind Extended Treatment(20weeks)
Arm/Group | Placebo IV | GSK2831781 450 mg IV | GSK2831781 300 mg IV | GSK2831781 150 mg IV | GSK2831781 45 mg IV | Placebo SC | GSK2831781 300 mg SC | Open-label GSK2831781 450 mg IV | Open-label GSK2831781 300 mg SC
Started | 0 | 0 | 0 | 0 | 0 | 5 | 8 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Period: Open-label Induction Phase (10 Weeks)
Arm/Group | Placebo IV | GSK2831781 450 mg IV | GSK2831781 300 mg IV | GSK2831781 150 mg IV | GSK2831781 45 mg IV | Placebo SC | GSK2831781 300 mg SC | Open-label GSK2831781 450 mg IV | Open-label GSK2831781 300 mg SC
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 42 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 30 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0
Period: Open-label Extended Treatment (20 Weeks)
Arm/Group | Placebo IV | GSK2831781 450 mg IV | GSK2831781 300 mg IV | GSK2831781 150 mg IV | GSK2831781 45 mg IV | Placebo SC | GSK2831781 300 mg SC | Open-label GSK2831781 450 mg IV | Open-label GSK2831781 300 mg SC
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Placebo IV: Participants were administered placebo via the intravenous (IV) route on Day 1, Weeks 2, 6 and 10. At Week 10, participants underwent Induction assessment including endoscopy.Participants were administered placebo via the intravenous (IV) route on Day 1, Weeks 2, 6 and 10. At Week 10, participants underwent Induction assessment including endoscopy.
- Total: Total of all reporting groups
Arm/Group | Placebo IV | GSK2831781 450 mg IV | GSK2831781 300 mg IV | GSK2831781 150 mg IV | GSK2831781 45 mg IV | Total
Number analyzed (Participants) | 27 | 48 | 11 | 10 | 8 | 104
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.9 (12.82) | 40.7 (12.70) | 37.6 (13.06) | 42.5 (15.06) | 40.6 (10.60) | 41.4 (12.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 22 | 4 | 4 | 1 | 43
  Male | 15 | 26 | 7 | 6 | 7 | 61
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian-Central/South Asian Heritage | 0 | 1 | 1 | 0 | 1 | 3
  Asian-East Asian Heritage | 2 | 0 | 0 | 0 | 0 | 2
  Asian-Japanese Heritage | 0 | 0 | 1 | 0 | 0 | 1
  Asian-South East Asian Heritage | 0 | 1 | 0 | 0 | 0 | 1
  White-Arabic/North African Heritage | 0 | 1 | 0 | 0 | 0 | 1
  White-White/Caucasian/European Heritage | 25 | 44 | 9 | 10 | 7 | 95
  Mixed White race | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)-Double-Blind Induction Phase
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; is a congenital anomaly/birth defect or other important medical events that may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed before. AEs and SAEs were collected up to Week 14 (for participants who later entered the Double Blind ETP) and Week 12 (for participants who later entered OL Induction Phase).
Time Frame: Up to a maximum of Week 14
Population: Safety Population comprised of all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo IV | GSK2831781 450 mg IV | GSK2831781 300 mg IV | GSK2831781 150 mg IV | GSK2831781 45 mg IV
Number analyzed (Participants) | 27 | 48 | 11 | 10 | 8
Participants
  AEs | 10 | 27 | 6 | 2 | 2
  SAEs | 0 | 6 | 1 | 0 | 0

2. Primary Outcome: Number of Participants With Worst-case Vital Signs Results by Potential Clinical Importance (PCI) Criteria Post-Baseline Relative to Baseline-Double-Blind Induction Phase
Description: Vital signs were measured in a seated or semi-supine position after 5 minutes rest. The clinical concern range for vital signs were: systolic blood pressure (SBP) (lower: <85 and upper: > 160 millimeters of mercury [mmHg]); diastolic blood pressure (DBP) (lower: <45 mmHg and upper: >100 mmHg); pulse rate (PR) (lower: <40 and upper: >110 beats per minute [bpm]) and temperature (Temp) (lower: <35 and upper: >38 degree Celsius). Participants were counted in the worst-case category that their value changed to (low, within range or no change, or high), unless there was no change in their category. Participants whose value category was unchanged (e.g. High to High), or whose value became within range, were recorded in the "To within (w/in) Range or No Change category". Participants were counted twice if the participant had values that changed "To Low" and "To High", so the percentages may not add to 100 percent (%).
Time Frame: Up to Week 10
Population: Safety Population. Only those participants with data available at the specified timepoints were analyzed (indicated by n=X in category titles)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo IV | GSK2831781 450 mg IV | GSK2831781 300 mg IV | GSK2831781 150 mg IV | GSK2831781 45 mg IV
Number analyzed (Participants) | 27 | 48 | 11 | 10 | 8
Participants
  DBP; To low; n=27, 47, 9, 8, 7: number analyzed (Participants) | 27 | 47 | 9 | 8 | 7
  DBP; To low; n=27, 47, 9, 8, 7 | 0 | 0 | 0 | 0 | 0
  DBP; To w/in range or no change; n=27, 47, 9, 8, 7: number analyzed (Participants) | 27 | 47 | 9 | 8 | 7
  DBP; To w/in range or no change; n=27, 47, 9, 8, 7 | 27 | 47 | 9 | 8 | 7
  DBP; To high; n=27, 47, 9, 8, 7: number analyzed (Participants) | 27 | 47 | 9 | 8 | 7
  DBP; To high; n=27, 47, 9, 8, 7 | 0 | 0 | 0 | 0 | 0
  SBP; To low; n=27, 47, 10, 9, 6: number analyzed (Participants) | 27 | 47 | 10 | 9 | 6
  SBP; To low; n=27, 47, 10, 9, 6 | 0 | 0 | 1 | 0 | 0
  SBP; To w/in range or no change; n=27, 47, 10, 9,6: number analyzed (Participants) | 27 | 47 | 10 | 9 | 6
  SBP; To w/in range or no change; n=27, 47, 10, 9,6 | 26 | 45 | 9 | 9 | 6
  SBP; To high; n=27, 47, 10, 9, 6: number analyzed (Participants) | 27 | 47 | 10 | 9 | 6
  SBP; To high; n=27, 47, 10, 9, 6 | 1 | 2 | 0 | 0 | 0
  PR; To low; n=27, 47, 11, 9, 8: number analyzed (Participants) | 27 | 47 | 11 | 9 | 8
  PR; To low; n=27, 47, 11, 9, 8 | 0 | 1 | 0 | 0 | 0
  PR; To w/in range or no change; n=27, 47, 11, 9, 8: number analyzed (Participants) | 27 | 47 | 11 | 9 | 8
  PR; To w/in range or no change; n=27, 47, 11, 9, 8 | 27 | 45 | 10 | 9 | 8
  PR; To high; n=27, 47, 11, 9, 8: number analyzed (Participants) | 27 | 47 | 11 | 9 | 8
  PR; To high; n=27, 47, 11, 9, 8 | 0 | 1 | 1 | 0 | 0
  Temp; To low; n=26, 46, 11, 10, 7: number analyzed (Participants) | 26 | 46 | 11 | 10 | 7
  Temp; To low; n=26, 46, 11, 10, 7 | 0 | 0 | 0 | 0 | 0
  Temp; To w/in range or no change; n=26,46,11,10,7: number analyzed (Participants) | 26 | 46 | 11 | 10 | 7
  Temp; To w/in range or no change; n=26,46,11,10,7 | 26 | 46 | 11 | 10 | 7
  Temp; To high; n=26, 46, 11, 10, 7: number analyzed (Participants) | 26 | 46 | 11 | 10 | 7
  Temp; To high; n=26, 46, 11, 10, 7 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Worst-case Hematology Results by PCI Criteria Post-Baseline Relative to Baseline-Double-Blind Induction Phase
Description: Blood samples were collected for the assessment of hematology parameters. The clinical concern range for the parameters were: hematocrit (Hct) (low: 0.201 and high: >0.599 proportion of red blood cells in blood); hemoglobin (Hgb) (low: <80 and high: >180 grams per liter [g/L]), lymphocytes (Lymph) (low: <0.8x10^9 cells/L); neutrophil (Neut) count (low: <1.5x10^9 cells/L); platelet (plat) count (low: <100x10^9 cells/L and high: >550x10^9 cells/L); leukocytes (leuko) (low: <3x10^9 cells/L and high: >20x10^9cells/L) and eosinophils (Eos) (high: >=1x10^9 cells/L). Participants were counted in the worst-case category that their value changed to (low, w/in range or no change, or high), unless there was no change in their category. Participants were counted twice if the participant had values that changed "To Low" and "To High", so the percentages may not add to 100%.
Time Frame: Up to Week 10
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo IV | GSK2831781 450 mg IV | GSK2831781 300 mg IV | GSK2831781 150 mg IV | GSK2831781 45 mg IV
Number analyzed (Participants) | 27 | 48 | 11 | 10 | 8
Participants
  Eos;w/in range or no change; n=25,45,9,8,7: number analyzed (Participants) | 25 | 45 | 9 | 8 | 7
  Eos;w/in range or no change; n=25,45,9,8,7 | 24 | 44 | 9 | 8 | 7
  Eos; To high; n=25,45,9,8,7: number analyzed (Participants) | 25 | 45 | 9 | 8 | 7
  Eos; To high; n=25,45,9,8,7 | 1 | 1 | 0 | 0 | 0
  Hct; To low; n=24,43,7,6,7: number analyzed (Participants) | 24 | 43 | 7 | 6 | 7
  Hct; To low; n=24,43,7,6,7 | 0 | 0 | 0 | 0 | 0
  Hct; To w/in range or no change; n=24,43,7,6,7: number analyzed (Participants) | 24 | 43 | 7 | 6 | 7
  Hct; To w/in range or no change; n=24,43,7,6,7 | 24 | 43 | 7 | 6 | 7
  Hct; To high; n=24,43,7,6,7: number analyzed (Participants) | 24 | 43 | 7 | 6 | 7
  Hct; To high; n=24,43,7,6,7 | 0 | 0 | 0 | 0 | 0
  Hgb; To low; n=24,45,5,7,7: number analyzed (Participants) | 24 | 45 | 5 | 7 | 7
  Hgb; To low; n=24,45,5,7,7 | 0 | 0 | 1 | 1 | 0
  Hgb; To w/in range or no change; n=24,45,5,7,7: number analyzed (Participants) | 24 | 45 | 5 | 7 | 7
  Hgb; To w/in range or no change; n=24,45,5,7,7 | 24 | 45 | 4 | 6 | 7
  Hgb; To high; n=24,45,5,7,7: number analyzed (Participants) | 24 | 45 | 5 | 7 | 7
  Hgb; To high; n=24,45,5,7,7 | 0 | 0 | 0 | 0 | 0
  Leuko; To low; n=27,43,8,9,6: number analyzed (Participants) | 27 | 43 | 8 | 9 | 6
  Leuko; To low; n=27,43,8,9,6 | 0 | 2 | 0 | 1 | 0
  Leuko; To w/in range or no change; n=27,43,8,9,6: number analyzed (Participants) | 27 | 43 | 8 | 9 | 6
  Leuko; To w/in range or no change; n=27,43,8,9,6 | 27 | 41 | 8 | 8 | 6
  Leuko; To high; n=27,43,8,9,6: number analyzed (Participants) | 27 | 43 | 8 | 9 | 6
  Leuko; To high; n=27,43,8,9,6 | 0 | 0 | 0 | 0 | 0
  Lymph; To low; n=26,45,8,8,8: number analyzed (Participants) | 26 | 45 | 8 | 8 | 8
  Lymph; To low; n=26,45,8,8,8 | 1 | 6 | 1 | 3 | 2
  Lymph; To w/in range or no change; n=26,45,8,8,8: number analyzed (Participants) | 26 | 45 | 8 | 8 | 8
  Lymph; To w/in range or no change; n=26,45,8,8,8 | 25 | 39 | 7 | 5 | 6
  Neut; To low; n=26,42,7,9,8: number analyzed (Participants) | 26 | 42 | 7 | 9 | 8
  Neut; To low; n=26,42,7,9,8 | 0 | 2 | 0 | 0 | 0
  Neut; To w/in range or no change; n=26,42,7,9,8: number analyzed (Participants) | 26 | 42 | 7 | 9 | 8
  Neut; To w/in range or no change; n=26,42,7,9,8 | 26 | 40 | 7 | 9 | 8
  Plat; To low; n=26,43,9,8,6: number analyzed (Participants) | 26 | 43 | 9 | 8 | 6
  Plat; To low; n=26,43,9,8,6 | 0 | 0 | 0 | 0 | 0
  Plat; To w/in range or no change; n=26,43,9,8,6: number analyzed (Participants) | 26 | 43 | 9 | 8 | 6
  Plat; To w/in range or no change; n=26,43,9,8,6 | 25 | 41 | 9 | 7 | 6
  Plat; To high; n=26,43,9,8,6: number analyzed (Participants) | 26 | 43 | 9 | 8 | 6
  Plat; To high; n=26,43,9,8,6 | 1 | 2 | 0 | 1 | 0

4. Primary Outcome: Number of Participants With Worst-case Clinical Chemistry Results by PCI Criteria Post-Baseline Relative to Baseline-Double-Blind Induction Phase
Description: Blood samples were collected for the assessment of clinical chemistry parameters. The clinical concern range for the parameters were: albumin (Alb) (low: <30 and high: >55 g/L), calcium (Ca) (low: 2 and high: 2.75 millimoles per liter [mmol/L]), urea (high: >10.5 mmol/L); creatinine (Creat) (high: change from Baseline >26 micromoles per liter [µmol/L]), glucose (Glu) (low: <3.5 and high: >7.9 mmol/L); estimated glomerular filtration rate (eGFR) (low: <60 milliliters per minute per 1.73 square meter [mL/min/1.73m^2)]; potassium (Pot) (low: <3 and high: >5.5 mmol/L); sodium (Sod) (low: <130 and high: >150 mmol/L); protein (Pro) (low: <50 and high: >85 g/L) and C-reactive protein (CRP) (high: >30 milligrams/L). Participants were counted in the worst-case category that their value changed to (low, w/in range or no change, or high), unless there was no change in their category.
Time Frame: Up to Week 10
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo IV | GSK2831781 450 mg IV | GSK2831781 300 mg IV | GSK2831781 150 mg IV | GSK2831781 45 mg IV
Number analyzed (Participants) | 27 | 48 | 11 | 10 | 8
Participants
  Alb; To low; n=26,42,7,6,6: number analyzed (Participants) | 26 | 42 | 7 | 6 | 6
  Alb; To low; n=26,42,7,6,6 | 0 | 2 | 0 | 1 | 0
  Alb; To w/in range or no change; n=26,42,7,6,6: number analyzed (Participants) | 26 | 42 | 7 | 6 | 6
  Alb; To w/in range or no change; n=26,42,7,6,6 | 26 | 40 | 7 | 5 | 6
  Alb; To high; n=26,42,7,6,6: number analyzed (Participants) | 26 | 42 | 7 | 6 | 6
  Alb; To high; n=26,42,7,6,6 | 0 | 0 | 0 | 0 | 0
  CRP; To w/in range or no change; n=26, 46,9,10,8: number analyzed (Participants) | 26 | 46 | 9 | 10 | 8
  CRP; To w/in range or no change; n=26, 46,9,10,8 | 25 | 36 | 7 | 9 | 8
  CRP; To high; n=26, 46,9,10,8: number analyzed (Participants) | 26 | 46 | 9 | 10 | 8
  CRP; To high; n=26, 46,9,10,8 | 1 | 10 | 2 | 1 | 0
  Cal; To low; n=26,45,7,4,7: number analyzed (Participants) | 26 | 45 | 7 | 4 | 7
  Cal; To low; n=26,45,7,4,7 | 1 | 0 | 0 | 1 | 0
  Cal; To w/in range or no change; n=26,45,7,4,7: number analyzed (Participants) | 26 | 45 | 7 | 4 | 7
  Cal; To w/in range or no change; n=26,45,7,4,7 | 25 | 45 | 7 | 3 | 7
  Cal; To high; n=26,45,7,4,7: number analyzed (Participants) | 26 | 45 | 7 | 4 | 7
  Cal; To high; n=26,45,7,4,7 | 0 | 0 | 0 | 0 | 0
  eGFR; To low; n=24,46,6,9,7: number analyzed (Participants) | 24 | 46 | 6 | 9 | 7
  eGFR; To low; n=24,46,6,9,7 | 1 | 1 | 0 | 1 | 0
  eGFR; To w/in range or no change; n=24,46,6,9,7: number analyzed (Participants) | 24 | 46 | 6 | 9 | 7
  eGFR; To w/in range or no change; n=24,46,6,9,7 | 23 | 45 | 6 | 8 | 7
  Glu; To low; n=26,45,5,8,7: number analyzed (Participants) | 26 | 45 | 5 | 8 | 7
  Glu; To low; n=26,45,5,8,7 | 1 | 1 | 0 | 0 | 0
  Glu; To w/in range or no change; n=26,45,5,8,7: number analyzed (Participants) | 26 | 45 | 5 | 8 | 7
  Glu; To w/in range or no change; n=26,45,5,8,7 | 25 | 43 | 5 | 8 | 7
  Glu; To high; n=26,45,5,8,7: number analyzed (Participants) | 26 | 45 | 5 | 8 | 7
  Glu; To high; n=26,45,5,8,7 | 0 | 1 | 0 | 0 | 0
  Pot; To low; n=27,44,10,7,8: number analyzed (Participants) | 27 | 44 | 10 | 7 | 8
  Pot; To low; n=27,44,10,7,8 | 0 | 1 | 0 | 0 | 0
  Pot; To w/in range or no change; n=27,44,10,7,8: number analyzed (Participants) | 27 | 44 | 10 | 7 | 8
  Pot; To w/in range or no change; n=27,44,10,7,8 | 27 | 43 | 10 | 7 | 8
  Pot; To high; n=27,44,10,7,8: number analyzed (Participants) | 27 | 44 | 10 | 7 | 8
  Pot; To high; n=27,44,10,7,8 | 0 | 0 | 0 | 0 | 0
  Pro; To low; n=26,43,7,5,7: number analyzed (Participants) | 26 | 43 | 7 | 5 | 7
  Pro; To low; n=26,43,7,5,7 | 0 | 0 | 0 | 0 | 0
  Pro To w/in range or no change; n=26,43,7,5,7: number analyzed (Participants) | 26 | 43 | 7 | 5 | 7
  Pro To w/in range or no change; n=26,43,7,5,7 | 26 | 41 | 7 | 5 | 7
  Pro; To high; n=26,43,7,5,7: number analyzed (Participants) | 26 | 43 | 7 | 5 | 7
  Pro; To high; n=26,43,7,5,7 | 0 | 2 | 0 | 0 | 0
  Sod; To low; n=25,45,10,8,8: number analyzed (Participants) | 25 | 45 | 10 | 8 | 8
  Sod; To low; n=25,45,10,8,8 | 0 | 0 | 0 | 0 | 0
  Sod; To w/in range or no change; n=25,45,10,8,8: number analyzed (Participants) | 25 | 45 | 10 | 8 | 8
  Sod; To w/in range or no change; n=25,45,10,8,8 | 25 | 45 | 10 | 8 | 8
  Sod; To high; n=25,45,10,8,8: number analyzed (Participants) | 25 | 45 | 10 | 8 | 8
  Sod; To high; n=25,45,10,8,8 | 0 | 0 | 0 | 0 | 0
  Urea; To w/in range or no change; n=26,45,5,6,7: number analyzed (Participants) | 26 | 45 | 5 | 6 | 7
  Urea; To w/in range or no change; n=26,45,5,6,7 | 26 | 45 | 5 | 6 | 7
  Urea; To high; n=26,45,5,6,7: number analyzed (Participants) | 26 | 45 | 5 | 6 | 7
  Urea; To high; n=26,45,5,6,7 | 0 | 0 | 0 | 0 | 0
  Creat; To w/in range or no change; n=27,44,9,6,7: number analyzed (Participants) | 27 | 44 | 9 | 6 | 7
  Creat; To w/in range or no change; n=27,44,9,6,7 | 27 | 44 | 9 | 6 | 7
  Creat; To high; n=27,44,9,6,7: number analyzed (Participants) | 27 | 44 | 9 | 6 | 7
  Creat; To high; n=27,44,9,6,7 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Worst-case Liver Function Results by PCI Criteria Post-Baseline Relative to Baseline-Double-Blind Induction Phase
Description: Blood samples were collected for the assessment of liver function parameters. The clinical concern range for liver function parameters were: alanine aminotransferase (ALT) (high: >=2 times upper limit of normal [ULN]); aspartate aminotransferase (AST) (high: >=2 times ULN); alkaline phosphatase (ALP) (high: >=2 times ULN) and bilirubin (Bil) (high: >=1.5 times ULN). Participants were counted in the worst-case category that their value changed to (within range or no change, or high), unless there was no change in their category. Participants whose value category was unchanged (e.g. High to High), or whose value became within range, were recorded in the "To within (w/in) Range or No Change category".
Time Frame: Up to Week 10
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo IV | GSK2831781 450 mg IV | GSK2831781 300 mg IV | GSK2831781 150 mg IV | GSK2831781 45 mg IV
Number analyzed (Participants) | 27 | 48 | 11 | 10 | 8
Participants
  ALT; To low; n=26,44,7,7,8: number analyzed (Participants) | 26 | 44 | 7 | 7 | 8
  ALT; To low; n=26,44,7,7,8 | 0 | 0 | 0 | 0 | 0
  ALT;To w/in range or no change; n=26,44,7,7,8: number analyzed (Participants) | 26 | 44 | 7 | 7 | 8
  ALT;To w/in range or no change; n=26,44,7,7,8 | 25 | 42 | 7 | 7 | 8
  ALT; To high; n=26,44,7,7,8: number analyzed (Participants) | 26 | 44 | 7 | 7 | 8
  ALT; To high; n=26,44,7,7,8 | 1 | 2 | 0 | 0 | 0
  AST; To low; n=26,45,7,8,7: number analyzed (Participants) | 26 | 45 | 7 | 8 | 7
  AST; To low; n=26,45,7,8,7 | 0 | 0 | 0 | 0 | 0
  AST; To w/in range or no change; n=26,45,7,8,7: number analyzed (Participants) | 26 | 45 | 7 | 8 | 7
  AST; To w/in range or no change; n=26,45,7,8,7 | 26 | 44 | 7 | 8 | 7
  AST; To high;n=26,45,7,8,7: number analyzed (Participants) | 26 | 45 | 7 | 8 | 7
  AST; To high;n=26,45,7,8,7 | 0 | 1 | 0 | 0 | 0
  ALP; To low; n=27,44,9,9,8: number analyzed (Participants) | 27 | 44 | 9 | 9 | 8
  ALP; To low; n=27,44,9,9,8 | 0 | 0 | 0 | 0 | 0
  ALP; To w/in range or no change; n=27,44,9,9,8: number analyzed (Participants) | 27 | 44 | 9 | 9 | 8
  ALP; To w/in range or no change; n=27,44,9,9,8 | 27 | 44 | 9 | 9 | 8
  ALP; To high; n=27,44,9,9,8: number analyzed (Participants) | 27 | 44 | 9 | 9 | 8
  ALP; To high; n=27,44,9,9,8 | 0 | 0 | 0 | 0 | 0
  Bil; To low; n=25,45,9,8,8: number analyzed (Participants) | 25 | 45 | 9 | 8 | 8
  Bil; To low; n=25,45,9,8,8 | 0 | 0 | 0 | 0 | 0
  Bil; To w/in range or no change; n=25,45,9,8,8: number analyzed (Participants) | 25 | 45 | 9 | 8 | 8
  Bil; To w/in range or no change; n=25,45,9,8,8 | 25 | 45 | 9 | 8 | 8
  Bil; To high; n=25,45,9,8,8: number analyzed (Participants) | 25 | 45 | 9 | 8 | 8
  Bil; To high; n=25,45,9,8,8 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Worst-case Urinalysis Results by PCI Criteria Post-Baseline Relative to Baseline-Double-Blind Induction Phase
Description: Urine samples were collected for the assessment of urine parameters by dipstick and microscopy. The dipstick test gives results in a semi-quantitative manner, and results can be read as Trace, 1+, 2+ indicating proportional concentrations in the urine sample. The clinical concern range for urine parameters were: Bil (high: >1+), glu (high: >1+); ketone (ket) (high: >2+); leuko (high: >1+); leukocyte esterase (LE); nitrite (nit) (high: positive); occult blood (OB) (high: >1+); potential of hydrogen (pH) (low: <4.6 and high: >8); prot (high:>1+); erythrocytes (erythro) (high: >3 cells per high power field [hpf]); specific gravity (sp gra) (low: <1.001 and high: >1.035) and urobilinogen (uro) (high: >1 mg/deciliter).
Time Frame: Up to Week 10
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo IV | GSK2831781 450 mg IV | GSK2831781 300 mg IV | GSK2831781 150 mg IV | GSK2831781 45 mg IV
Number analyzed (Participants) | 27 | 48 | 11 | 10 | 8
Participants
  Bil; To w/in range or no change; n=27,47,10,9,8: number analyzed (Participants) | 27 | 47 | 10 | 9 | 8
  Bil; To w/in range or no change; n=27,47,10,9,8 | 27 | 46 | 10 | 9 | 8
  Bil; To high; n=27,47,10,9,8: number analyzed (Participants) | 27 | 47 | 10 | 9 | 8
  Bil; To high; n=27,47,10,9,8 | 0 | 1 | 0 | 0 | 0
  Glu; To w/in range or no change; n=27,47,10,10,8: number analyzed (Participants) | 27 | 47 | 10 | 10 | 8
  Glu; To w/in range or no change; n=27,47,10,10,8 | 27 | 47 | 10 | 10 | 8
  Glu; To high; n=27,47,10,10,8: number analyzed (Participants) | 27 | 47 | 10 | 10 | 8
  Glu; To high; n=27,47,10,10,8 | 0 | 0 | 0 | 0 | 0
  Ket; To w/in range or no change; n=27,47,10,8,8: number analyzed (Participants) | 27 | 47 | 10 | 8 | 8
  Ket; To w/in range or no change; n=27,47,10,8,8 | 25 | 47 | 10 | 7 | 8
  Ket; To high; n=27,47,10,8,8: number analyzed (Participants) | 27 | 47 | 10 | 8 | 8
  Ket; To high; n=27,47,10,8,8 | 2 | 0 | 0 | 1 | 0
  LE; To w/in range or no change; n=26,45,9,8,8: number analyzed (Participants) | 26 | 45 | 9 | 8 | 8
  LE; To w/in range or no change; n=26,45,9,8,8 | 25 | 37 | 9 | 8 | 8
  LE; To high; n=26,45,9,8,8: number analyzed (Participants) | 26 | 45 | 9 | 8 | 8
  LE; To high; n=26,45,9,8,8 | 1 | 8 | 0 | 0 | 0
  Nit; To w/in range or no change; n=27,47,10,10,8: number analyzed (Participants) | 27 | 47 | 10 | 10 | 8
  Nit; To w/in range or no change; n=27,47,10,10,8 | 27 | 44 | 9 | 8 | 8
  Nit; To high; n=27,47,10,10,8: number analyzed (Participants) | 27 | 47 | 10 | 10 | 8
  Nit; To high; n=27,47,10,10,8 | 0 | 3 | 1 | 2 | 0
  OB; To w/in range or no change; n=26,46,9,10,8: number analyzed (Participants) | 26 | 46 | 9 | 10 | 8
  OB; To w/in range or no change; n=26,46,9,10,8 | 24 | 42 | 9 | 10 | 8
  OB; To high; n=26,46,9,10,8: number analyzed (Participants) | 26 | 46 | 9 | 10 | 8
  OB; To high; n=26,46,9,10,8 | 2 | 4 | 0 | 0 | 0
  pH; To low; n=27,46,9,10,7: number analyzed (Participants) | 27 | 46 | 9 | 10 | 7
  pH; To low; n=27,46,9,10,7 | 0 | 0 | 0 | 0 | 0
  pH; To w/in range or no change; n=27,46,9,10,7: number analyzed (Participants) | 27 | 46 | 9 | 10 | 7
  pH; To w/in range or no change; n=27,46,9,10,7 | 26 | 46 | 9 | 10 | 7
  pH; To high; n=27,46,9,10,7: number analyzed (Participants) | 27 | 46 | 9 | 10 | 7
  pH; To high; n=27,46,9,10,7 | 1 | 0 | 0 | 0 | 0
  Prot; To w/in range or no change; n=25,47,10,9,8: number analyzed (Participants) | 25 | 47 | 10 | 9 | 8
  Prot; To w/in range or no change; n=25,47,10,9,8 | 24 | 43 | 10 | 9 | 8
  Prot; To high; n=25,47,10,9,8: number analyzed (Participants) | 25 | 47 | 10 | 9 | 8
  Prot; To high; n=25,47,10,9,8 | 1 | 4 | 0 | 0 | 0
  Uro; To w/in range or no change; n=27,47,10,8,8: number analyzed (Participants) | 27 | 47 | 10 | 8 | 8
  Uro; To w/in range or no change; n=27,47,10,8,8 | 27 | 47 | 10 | 8 | 8
  Uro; To high; n=27,47,10,8,8: number analyzed (Participants) | 27 | 47 | 10 | 8 | 8
  Uro; To high; n=27,47,10,8,8 | 0 | 0 | 0 | 0 | 0
  Leuko; To w/in range or no change; n=9,18,2,3,1: number analyzed (Participants) | 9 | 18 | 2 | 3 | 1
  Leuko; To w/in range or no change; n=9,18,2,3,1 | 8 | 15 | 1 | 3 | 1
  Leuko; To high; n=9,18,2,3,1: number analyzed (Participants) | 9 | 18 | 2 | 3 | 1
  Leuko; To high; n=9,18,2,3,1 | 1 | 3 | 1 | 0 | 0
  Erythro; To w/in range or no change; n=9,18,2,3,1: number analyzed (Participants) | 9 | 18 | 2 | 3 | 1
  Erythro; To w/in range or no change; n=9,18,2,3,1 | 9 | 16 | 1 | 3 | 1
  Erythro; To high; n=9,18,2,3,1: number analyzed (Participants) | 9 | 18 | 2 | 3 | 1
  Erythro; To high; n=9,18,2,3,1 | 0 | 2 | 1 | 0 | 0
  Sp gra; To low; n=25,47,5,7,8: number analyzed (Participants) | 25 | 47 | 5 | 7 | 8
  Sp gra; To low; n=25,47,5,7,8 | 0 | 0 | 0 | 0 | 0
  Sp gra; To w/in range or no change; n=25,47,5,7,8: number analyzed (Participants) | 25 | 47 | 5 | 7 | 8
  Sp gra; To w/in range or no change; n=25,47,5,7,8 | 21 | 44 | 5 | 7 | 8
  Sp gra; To high; n=25,47,5,7,8: number analyzed (Participants) | 25 | 47 | 5 | 7 | 8
  Sp gra; To high; n=25,47,5,7,8 | 4 | 3 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Maximum Corrected QT (QTc) Values Post-Baseline Relative to Baseline-Double-Blind Induction Phase
Description: Twelve lead electrocardiograms (ECGs) were obtained using an ECG machine that automatically calculated the QT interval corrected for heart rate according to either Bazett's formula (QTcB) or Fridericia's formula (QTcF). The clinical concern range for the QTcB and QTcF intervals was upper: >450 milliseconds.
Time Frame: Up to Week 10
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo IV | GSK2831781 450 mg IV | GSK2831781 300 mg IV | GSK2831781 150 mg IV | GSK2831781 45 mg IV
Number analyzed (Participants) | 27 | 48 | 11 | 10 | 8
Participants
  QTcB; No change or decrease to <450; n=26,44,8,9,7: number analyzed (Participants) | 26 | 44 | 8 | 9 | 7
  QTcB; No change or decrease to <450; n=26,44,8,9,7 | 22 | 41 | 6 | 7 | 7
  QTcB; Any increase to >=450; n=26,44,8,9,7: number analyzed (Participants) | 26 | 44 | 8 | 9 | 7
  QTcB; Any increase to >=450; n=26,44,8,9,7 | 4 | 3 | 2 | 2 | 0
  QTcF; No change or decrease to <450; n=26,46,7,9,7: number analyzed (Participants) | 26 | 46 | 7 | 9 | 7
  QTcF; No change or decrease to <450; n=26,46,7,9,7 | 26 | 45 | 7 | 8 | 7
  QTcF; Any increase to >=450; n=26,46,7,9,7: number analyzed (Participants) | 26 | 46 | 7 | 9 | 7
  QTcF; Any increase to >=450; n=26,46,7,9,7 | 0 | 1 | 0 | 1 | 0

8. Primary Outcome: Change From Baseline in Complete 4-domain Mayo Score at Week 10
Description: The Complete 4-domain Mayo Score is a 12-point scoring system where disease is evaluated based on the four components: stool frequency, rectal bleeding, physician global assessment (PGA) and endoscopic appearance (with mild friability associated with an endoscopic score of 1). The score for each component ranges from 0 (normal/none) to 3 (severe). The complete Mayo score is calculated as the sum of four components and ranges from 0 to 12. Higher scores indicate greater disease severity. Baseline value was the latest pre-dose assessment with a non-missing value from Double-Blind Induction study phase. Change from Baseline was calculated as value at specified time point minus Baseline value.
Time Frame: Baseline and Week 10
Population: Intent-To-Treat-Exposed (ITTE) Population comprised of all enrolled participants who received at least one dose of study treatment, and who had at least one valid post dose assessment. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo IV | GSK2831781 450 mg IV | GSK2831781 300 mg IV | GSK2831781 150 mg IV | GSK2831781 45 mg IV
Number analyzed (Participants) | 21 | 36 | 4 | 2 | 3
Scores on a scale | -1.5 (0.45) | -1.4 (0.36) | -0.3 (0.48) | -1.0 (2.00) | -2.3 (0.33)

9. Secondary Outcome: Number of Participants With AEs and SAEs-Double-Blind Extended Treatment Phase
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; is a congenital anomaly/birth defect or other important medical events that may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed before.
Time Frame: Week 14 to 30
Population: Safety Extended Treatment Population comprised of all participants who received at least one dose of study treatment in the Extended Treatment Phase
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo SC | GSK2831781 300 mg SC
Number analyzed (Participants) | 5 | 8
Participants
  AEs | 1 | 3
  SAEs | 0 | 1

10. Secondary Outcome: Number of Participants With Worst-case Vital Signs Results by PCI Criteria Post-Baseline Relative to Baseline-Double-Blind Extended Treatment Phase
Description: Vital signs were measured in a seated or semi-supine position after 5 minutes rest. The clinical concern range for vital signs were: SBP (lower: <85 and upper: > 160 mmHg); DBP (lower: <45 mmHg and upper: >100 mmHg); PR (lower: <40 and upper: >110 bpm) and Temp (lower: <35 and upper: >38 degree Celsius). Participants were counted in the worst-case category that their value changed to (low, within range or no change, or high), unless there was no change in their category. Participants whose value category was unchanged (e.g. High to High), or whose value became within range, were recorded in the "To w/in Range or No Change category". Participants were counted twice if the participant had values that changed "To Low" and "To High", so the percentages may not add to 100%.
Time Frame: Week 14 to 30
Population: Safety Extended Treatment Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo SC | GSK2831781 300 mg SC
Number analyzed (Participants) | 5 | 8
Participants
  DBP; To low | 0 | 0
  DBP; To w/in range or no change | 5 | 8
  DBP; To high | 0 | 0
  SBP; To low | 0 | 0
  SBP; To w/in range or no change | 5 | 8
  SBP; To high | 0 | 0
  PR; To low | 0 | 0
  PR; To w/in range or no change | 5 | 8
  PR; To high | 0 | 0
  Temp; To low | 0 | 0
  Temp; To w/in range or no change | 5 | 8
  Temp; To high | 0 | 0

11. Secondary Outcome: Number of Participants With Worst-case Hematology Results by PCI Criteria Post-Baseline Relative to Baseline-Double-Blind Extended Treatment Phase
Description: Blood samples were collected for the assessment of hematology parameters. The clinical concern range for the parameters were: Hct (low: 0.201 and high: >0.599 proportion of red blood cells in blood); Hgb (low: <80 and high: >180 g/L), Lymph (low: <0.8x10^9 cells/L); Neut count (low: <1.5x10^9 cells/L); plat count (low: <100x10^9 cells/L and high: >550x10^9 cells/L); leuko (low: <3x10^9 cells/L and high: >20x10^9cells/L) and Eos (high: >=1x10^9 cells/L). Participants were counted in the worst-case category that their value changed to (low, within range or no change, or high), unless there was no change in their category. Participants whose value category was unchanged (e.g. High to High), or whose value became within range, were recorded in the "To w/in Range or No Change category". Participants were counted twice if the participant had values that changed "To Low" and "To High", so the percentages may not add to 100%.
Time Frame: Week 14 to 30
Population: Safety Extended Treatment Population. Only those participants with data available at the specified timepoints were analyzed (indicated by n=X in category titles)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo SC | GSK2831781 300 mg SC
Number analyzed (Participants) | 5 | 8
Participants
  Eos;To w/in range or no change; n=4,8: number analyzed (Participants) | 4 | 8
  Eos;To w/in range or no change; n=4,8 | 4 | 8
  Eos; To high; n=4,8: number analyzed (Participants) | 4 | 8
  Eos; To high; n=4,8 | 0 | 0
  Hct; To low; n=5,8 | 0 | 0
  Hct; To w/in range or no change; n=5,8 | 5 | 8
  Hct; To high; n=5,8 | 0 | 0
  Hgb; To low; n=5,8 | 0 | 0
  Hgb; To w/in range or no change; n=5,8 | 5 | 8
  Hgb; To high; n=5,8 | 0 | 0
  Leuko; To low; n=5,8 | 0 | 0
  Leuko; To w/in range or no change; n=5,8 | 5 | 8
  Leuko; To high; n=5,8 | 0 | 0
  Lymph; To low; n=5,8 | 0 | 2
  Lymph; To w/in range or no change; n=5,8 | 5 | 6
  Neut; To low; n=5,8 | 0 | 0
  Neut; To w/in range or no change; n=5,8 | 5 | 8
  Plat; To low; n=5,8 | 0 | 0
  Plat; To w/in range or no change; n=5,8 | 5 | 6
  Plat; To high; n=5,8 | 0 | 2

12. Secondary Outcome: Number of Participants With Worst-case Clinical Chemistry Results by PCI Criteria Post-Baseline Relative to Baseline-Double-Blind Extended Treatment Phase
Description: Blood samples were collected for the assessment of clinical chemistry parameters. The clinical concern range for the parameters were: Alb (low: <30 and high: >55 g/L), C) (low: 2 and high: 2.75 mmol/L), urea (high: >10.5 mmol/L); Creat (high: change from Baseline >26 µmol/L), Glu (low: <3.5 and high: >7.9 mmol/L); eGFR (low: <60 mL/min/1.73m^2]; Pot low: <3 and high: >5.5 mmol/L); Sod (low: <130 and high: >150 mmol/L); Pro (low: <50 and high: >85 g/L) and CRP (high: >30 milligrams/L). Participants were counted in the worst-case category that their value changed to (low, within range or no change, or high), unless there was no change in their category. Participants whose value category was unchanged (e.g. High to High), or whose value became within range, were recorded in the "To w/in Range or No Change category". Participants were counted twice if the participant had values that changed "To Low" and "To High", so the percentages may not add to 100%.
Time Frame: Week 14 to 30
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo SC | GSK2831781 300 mg SC
Number analyzed (Participants) | 5 | 8
Participants
  Alb; To low; n=5,8 | 0 | 1
  Alb; To w/in range or no change; n=5,8 | 5 | 7
  Alb; To high; n=5,8 | 0 | 0
  CRP; To w/in range or no change; n=5,8 | 5 | 6
  CRP; To high; n=5,8 | 0 | 2
  Cal; To low; n=5,8 | 0 | 0
  Cal; To w/in range or no change; n=5,8 | 5 | 8
  Cal; To high; n=5,8 | 0 | 0
  eGFR; To low; n=4,8: number analyzed (Participants) | 4 | 8
  eGFR; To low; n=4,8 | 0 | 1
  eGFR; To w/in range or no change; n=4,8: number analyzed (Participants) | 4 | 8
  eGFR; To w/in range or no change; n=4,8 | 4 | 7
  Glu; To low; n=5,8 | 0 | 0
  Glu; To w/in range or no change; n=5,8 | 5 | 8
  Glu; To high; n=5,8 | 0 | 0
  Pot; To low;n=4,8: number analyzed (Participants) | 4 | 8
  Pot; To low;n=4,8 | 0 | 0
  Pot; To w/in range or no change; n=4,8: number analyzed (Participants) | 4 | 8
  Pot; To w/in range or no change; n=4,8 | 4 | 8
  Pot; To high; n=4,8: number analyzed (Participants) | 4 | 8
  Pot; To high; n=4,8 | 0 | 0
  Pro; To low; n=5,8 | 0 | 0
  Pro To w/in range or no change; n=5,8 | 5 | 8
  Pro; To high; n=5,8 | 0 | 0
  Sod; To low; n=4,8: number analyzed (Participants) | 4 | 8
  Sod; To low; n=4,8 | 0 | 0
  Sod; To w/in range or no change; n=4,8: number analyzed (Participants) | 4 | 8
  Sod; To w/in range or no change; n=4,8 | 4 | 8
  Sod; To high; n=4,8: number analyzed (Participants) | 4 | 8
  Sod; To high; n=4,8 | 0 | 0
  Urea; To w/in range or no change; n=5,8 | 5 | 8
  Urea; To high; n=5,8 | 0 | 0
  Creat; To w/in range or no change; n=5,8 | 5 | 8
  Creat; To high; n=5,8 | 0 | 0

13. Secondary Outcome: Number of Participants With Worst-case Liver Function Results by PCI Criteria Post-Baseline Relative to Baseline-Double-Blind Extended Treatment Phase
Description: Blood samples were collected for the assessment of liver function parameters. The clinical concern range for liver function parameters were: ALT (high: >=2 times ULN); AST (high: >=2 times ULN); ALP (high: >=2 times ULN) and Bil (high: >=1.5 times ULN). Participants were counted in the worst-case category that their value changed to (low, within range or no change, or high), unless there was no change in their category. Participants whose value category was unchanged (e.g. High to High), or whose value became within range, were recorded in the "To w/in Range or No Change category".
Time Frame: Week 14 to 30
Population: Safety Extended Treatment Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo SC | GSK2831781 300 mg SC
Number analyzed (Participants) | 5 | 8
Participants
  ALT; To low | 0 | 0
  ALT;To w/in range or no change | 5 | 8
  ALT; To high | 0 | 0
  AST; To low | 0 | 0
  AST; To w/in range or no change | 5 | 8
  AST; To high | 0 | 0
  ALP; To low | 0 | 0
  ALP; To w/in range or no change | 5 | 8
  ALP; To high: number analyzed (Participants) | 4 | 8
  ALP; To high | 0 | 0
  Bil; To low: number analyzed (Participants) | 4 | 8
  Bil; To low | 0 | 0
  Bil; To w/in range or no change | 5 | 8
  Bil; To high | 0 | 0

14. Secondary Outcome: Number of Participants With Worst-case Urinalysis Results by PCI Criteria Post-Baseline Relative to Baseline-Double-Blind Extended Treatment Phase
Description: Urine samples were collected for the assessment of urine parameters by dipstick and microscopy. The dipstick test gives results in a semi-quantitative manner, and results can be read as Trace, 1+, 2+ indicating proportional concentrations in the urine sample. The clinical concern range for urine parameters were: Bil (high: >1+), glu (high: >1+); ket (high: >2+); leuko (high: >1+); LE; nit (high: positive); OB (high: >1+); pH (low: <4.6 and high: >8); prot (high:>1+); erythro (high: >3 cells per hpf); sp gra (low: <1.001 and high: >1.035) and uro (high: >1 mg/deciliter).
Time Frame: Week 14 to 30
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo SC | GSK2831781 300 mg SC
Number analyzed (Participants) | 5 | 8
Participants
  Bil; To w/in range or no change; n=5,8 | 5 | 8
  Bil; To high; n=5,8 | 0 | 0
  Glu; To w/in range or no change; n=5,8 | 5 | 8
  Glu; To high; n=5,8 | 0 | 0
  Ket; To w/in range or no change; n=5,8 | 5 | 8
  Ket; To high; n=5,8 | 0 | 0
  LE; To w/in range or no change; n=5,8 | 3 | 8
  LE; To high; n=5,8 | 2 | 0
  Nit; To w/in range or no change; n=5,8 | 5 | 7
  Nit; To high; n=5,8 | 0 | 1
  OB; To w/in range or no change; n=5,8 | 4 | 7
  OB; To high; n=5,8 | 1 | 1
  pH; To low; n=5,8 | 0 | 0
  pH; To w/in range or no change; n=5,8 | 5 | 8
  pH; To high; n=5,8 | 0 | 0
  Prot; To w/in range or no change; n=5,8 | 4 | 8
  Prot; To high; n=5,8 | 1 | 0
  Uro; To w/in range or no change; n=5,8 | 5 | 8
  Uro; To high; n=5,8 | 0 | 0
  Leuko; To w/in range or no change; n=1,2: number analyzed (Participants) | 1 | 2
  Leuko; To w/in range or no change; n=1,2 | 1 | 1
  Leuko; To high; n=1,2: number analyzed (Participants) | 1 | 2
  Leuko; To high; n=1,2 | 0 | 1
  Erythro; To w/in range or no change; n=1,2: number analyzed (Participants) | 1 | 2
  Erythro; To w/in range or no change; n=1,2 | 1 | 2
  Erythro; To high; n=1,2: number analyzed (Participants) | 1 | 2
  Erythro; To high; n=1,2 | 0 | 0
  Sp gra; To low; n=5,8 | 0 | 0
  Sp gra; To w/in range or no change; n=5,8 | 4 | 6
  Sp gra; To high; n=5,8 | 1 | 2

15. Secondary Outcome: Number of Participants With Maximum QTc Values Post-Baseline Relative to Baseline-Double-Blind Extended Treatment Phase
Description: Twelve lead ECGs were obtained using an ECG machine that automatically calculated the QTcB and QTcF intervals. The clinical concern range for the QTcB and QTcF intervals was upper: >450 milliseconds.
Time Frame: Week 14 to 30
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo SC | GSK2831781 300 mg SC
Number analyzed (Participants) | 4 | 8
Participants
  QTcB; No change or decrease to <450; n=4,6: number analyzed (Participants) | 4 | 6
  QTcB; No change or decrease to <450; n=4,6 | 4 | 6
  QTcB; Any increase to >=450; n=4,6: number analyzed (Participants) | 4 | 6
  QTcB; Any increase to >=450; n=4,6 | 0 | 0
  QTcF; No change or decrease to <450; n=3,6: number analyzed (Participants) | 3 | 6
  QTcF; No change or decrease to <450; n=3,6 | 3 | 6
  QTcF; Any increase to >=450; n=3,6: number analyzed (Participants) | 3 | 6
  QTcF; Any increase to >=450; n=3,6 | 0 | 0

16. Secondary Outcome: Number of Participants With Adapted Mayo Endoscopic Score of 0 or 1 at Week 10-Double-Blind Induction Phase
Description: The adapted Mayo clinical score consists of three components: stool frequency, rectal bleeding, and endoscopic appearance. The score for each component ranges from 0 (normal/none) to 3 (severe). The adapted Mayo endoscopic score of 0 indicates normal or inactive disease and 1 indicates mild disease (erythema, decreased vascular pattern).
Time Frame: Week 10
Population: ITTE Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo IV | GSK2831781 450 mg IV | GSK2831781 300 mg IV | GSK2831781 150 mg IV | GSK2831781 45 mg IV
Number analyzed (Participants) | 21 | 36 | 4 | 2 | 3
Participants | 4 | 3 | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With Adapted Mayo Clinical Remission at Week 10-Double-Blind Induction Phase
Description: The adapted Mayo clinical score is based on the complete 4-domain Mayo clinical score, but without the PGA. It consists of three components: stool frequency, rectal bleeding, and mucosal endoscopic appearance. The score for each component ranges from 0 (normal/none) to 3 (severe). The total adapted Mayo score is calculated as the sum of all three components and ranges from 0 to 9. Higher scores indicate greater disease severity. Clinical remission is defined as adapted Mayo Clinical Score of <=2 with no individual sub-score >1 and a rectal bleeding sub score of 0 with stool frequency sub score not greater than Baseline.
Time Frame: Week 10
Population: ITTE Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo IV | GSK2831781 450 mg IV | GSK2831781 300 mg IV | GSK2831781 150 mg IV | GSK2831781 45 mg IV
Number analyzed (Participants) | 21 | 36 | 4 | 2 | 3
Participants | 0 | 1 | 0 | 0 | 0

18. Secondary Outcome: Number of Participants With Adapted Mayo Clinical Response at Week 10-Double-Blind Induction Phase
Description: The adapted Mayo clinical score is based on the complete 4-domain Mayo clinical score, but without the PGA. It consists of three components: stool frequency, rectal bleeding, and mucosal endoscopic appearance. The score for each component ranges from 0 (normal/none) to 3 (severe). The total adapted Mayo score is calculated as the sum of all three components and ranges from 0 to 9. Higher scores indicate greater disease severity. Clinical response is defined as reduction in adapted Mayo clinical score >=3 points from Baseline and >=30% from Baseline and decrease in the rectal bleeding sub-score of >=1 point from Baseline (or a score of 0 or 1).
Time Frame: Week 10
Population: ITTE Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo IV | GSK2831781 450 mg IV | GSK2831781 300 mg IV | GSK2831781 150 mg IV | GSK2831781 45 mg IV
Number analyzed (Participants) | 21 | 36 | 4 | 2 | 3
Participants | 5 | 6 | 0 | 1 | 0

19. Secondary Outcome: Number of Participants With Symptomatic Remission at Week 10-Double-Blind Induction Phase
Description: The Complete 4-domain Mayo Score is a 12-point scoring system where disease is evaluated based on the four components: stool frequency, rectal bleeding, PGA and endoscopic appearance (with mild friability associated with an endoscopic score of 1). Symptomatic remission is defined as a rectal bleeding subscore of 0, and a stool frequency subscore of <=1, with no worsening from Baseline.
Time Frame: Week 10
Population: ITTE Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo IV | GSK2831781 450 mg IV | GSK2831781 300 mg IV | GSK2831781 150 mg IV | GSK2831781 45 mg IV
Number analyzed (Participants) | 21 | 36 | 4 | 2 | 3
Participants | 5 | 5 | 0 | 1 | 1

20. Secondary Outcome: Change From Baseline in Partial Mayo Score Over Time-Double-Blind Induction Phase
Description: The partial Mayo clinical score is based on the complete 4-domain Mayo clinical score but without the endoscopy sub-score. It consists of three components: stool frequency, rectal bleeding, and PGA. The score for each component ranges from 0 (normal/none) to 3 (severe). The total partial Mayo score is calculated as the sum of all three components and ranges from 0 to 9. Higher scores indicate greater disease severity. Baseline value was the latest pre-dose assessment with a non-missing value from Double-Blind Induction study phase. Change from Baseline was calculated as value at specified time point minus Baseline value.
Time Frame: Baseline and Weeks 2, 4, 6, and 10
Population: ITTE Population. Only those participants with data available at the specified time points were analyzed (indicated by n=X in category titles).
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo IV | GSK2831781 450 mg IV | GSK2831781 300 mg IV | GSK2831781 150 mg IV | GSK2831781 45 mg IV
Number analyzed (Participants) | 27 | 48 | 11 | 10 | 8
Scores on a scale
  Week 2; n=27, 47, 11, 10, 8: number analyzed (Participants) | 27 | 47 | 11 | 10 | 8
  Week 2; n=27, 47, 11, 10, 8 | -0.8 (0.33) | -0.6 (0.22) | -1.0 (0.50) | 0.5 (0.54) | -1.3 (0.65)
  Week 4; n=26, 46, 8, 8, 7: number analyzed (Participants) | 26 | 46 | 8 | 8 | 7
  Week 4; n=26, 46, 8, 8, 7 | -1.0 (0.31) | -0.7 (0.28) | -1.4 (0.60) | -0.4 (0.18) | -1.7 (0.52)
  Week 6; n=24, 44, 8, 6, 8: number analyzed (Participants) | 24 | 44 | 8 | 6 | 8
  Week 6; n=24, 44, 8, 6, 8 | -1.3 (0.40) | -0.8 (0.31) | -1.0 (0.53) | -0.8 (0.31) | -2.6 (0.53)
  Week 10; n=22, 39, 4, 4, 4: number analyzed (Participants) | 22 | 39 | 4 | 4 | 4
  Week 10; n=22, 39, 4, 4, 4 | -1.1 (0.44) | -1.0 (0.32) | 0.3 (0.48) | -1.0 (0.41) | -2.0 (0.41)

21. Secondary Outcome: Change From Baseline in Adapted Mayo Endoscopy Score at Week 10-Double-Blind Induction Phase
Description: The adapted Mayo clinical score is based on the complete 4-domain Mayo clinical score, but without the PGA. It consists of three components: stool frequency, rectal bleeding, and mucosal endoscopic appearance. The total adapted Mayo endoscopy score ranges from 0 (normal or inactive disease) to 3 (severe disease [spontaneous bleeding, ulceration]). Baseline value was the latest pre-dose assessment with a non-missing value from Double-Blind Induction study phase. Change from Baseline was calculated as value at specified time point minus Baseline value.
Time Frame: Baseline and Week 10
Population: ITTE Population. Only those participants with data available at the specified time points were analyzed
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo IV | GSK2831781 450 mg IV | GSK2831781 300 mg IV | GSK2831781 150 mg IV | GSK2831781 45 mg IV
Number analyzed (Participants) | 21 | 36 | 4 | 2 | 3
Scores on a scale | -0.2 (0.14) | -0.1 (0.12) | 0.0 (0.00) | 0.5 (0.50) | -0.3 (0.33)

22. Secondary Outcome: Change From Baseline in Ulcerative Colitis Endoscopic Index of Severity (UCEIS) at Week 10-Double-Blind Induction Phase
Description: UCEIS was used as an additional tool to assess disease activity based on 3 sub-scales: endoscopic vascular pattern, bleeding, erosions and ulcerations. Individual sub-scale scores were vascular pattern (0=Normal, 1=Patchy loss, 2=Obliterated); bleeding (0=None, 1=Mucosal, 2=Luminal mild, 3=Luminal severe); erosions and ulcerations (0=None, 1=Erosions, 2=Superficial ulcer, 3=Deep ulcer). UCEIS total score was calculated as the sum of all 3 sub-scale scores and ranges from 0 to 8, with higher scores indicating more severe disease. Baseline value was the latest pre-dose assessment with a non-missing value from Double-Blind Induction study phase. Change from Baseline was calculated as value at specified time point minus Baseline value.
Time Frame: Baseline and Week 10
Population: ITTE Population. Only those participants with data available at the specified time points were analyzed
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo IV | GSK2831781 450 mg IV | GSK2831781 300 mg IV | GSK2831781 150 mg IV | GSK2831781 45 mg IV
Number analyzed (Participants) | 21 | 36 | 4 | 2 | 3
Scores on a scale | -0.1 (0.41) | -0.0 (0.25) | 0.5 (0.65) | 1.0 (0.00) | 0.0 (0.58)

23. Secondary Outcome: Number of Responders for Robarts Histopathology Index (RHI) Remission at Week 10-Double-Blind Induction Phase
Description: RHI was assessed by central reading of gut pinch biopsies. The RHI Score is a continuous score, ranging from 0-33 with higher scores indicating more severe disease. RHI Remission is defined as an RHI score <=6. Responders were defined as number of participants with RHI score <=6.
Time Frame: Week 10
Population: ITTE Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo IV | GSK2831781 450 mg IV | GSK2831781 300 mg IV | GSK2831781 150 mg IV | GSK2831781 45 mg IV
Number analyzed (Participants) | 21 | 36 | 4 | 2 | 3
Participants | 4 | 5 | 0 | 0 | 0

24. Secondary Outcome: Number of Responders for Nancy Histological Index Remission at Week 10-Double-Blind Induction Phase
Description: Nancy Histological Index was assessed by central reading of gut pinch biopsies. Key domains for scoring of the indices include chronic inflammatory infiltrate, neutrophils in the epithelium, lamina propria neutrophils, erosion and ulceration scored from 0 to 3 and multiplied by a weighting factor. The total Nancy Histological Index score is calculated by summing the weighted scores of the histological items, with total scores ranging from 0 (no disease activity) to 33 (severe disease activity). Nancy Index Remission was defined as a grade of 0 or 1. Responders were defined as number of participants with Nancy Index score of 0 or 1.
Time Frame: Week 10
Population: ITTE Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo IV | GSK2831781 450 mg IV | GSK2831781 300 mg IV | GSK2831781 150 mg IV | GSK2831781 45 mg IV
Number analyzed (Participants) | 21 | 36 | 4 | 2 | 3
Participants | 4 | 4 | 0 | 0 | 0

25. Secondary Outcome: Number of Responders for Geboes Histological Index Remission at Week 10-Double-Blind Induction Phase
Description: The Geboes Index is divided in 6 grades: architectural changes [grade 0], chronic inflammatory infiltrate [grade 1], lamina propria neutrophils and eosinophils [grade 2], neutrophils in epithelium [grade 3], crypt destruction [grade 4] and erosions or ulcerations [grade 5]. The subscores for grade 0 to 4 ranges from 0 (none/no abnormality) to 3 (marked increase/severe abnormality) and for grade 5 ranges from 0 (No erosion, ulceration, or granulation tissue) to 4 (Ulcer or granulation tissue). The overall Geboes score is derived by summing the subscores of the grades and ranges from 0 to 22, with higher scores indicating greater disease severity. Geboes Histological Remission was defined as a Geboes score <2. Responders were defined as number of participants with Geboes score <2.
Time Frame: Week 10
Population: ITTE Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo IV | GSK2831781 450 mg IV | GSK2831781 300 mg IV | GSK2831781 150 mg IV | GSK2831781 45 mg IV
Number analyzed (Participants) | 21 | 36 | 4 | 2 | 3
Participants | 1 | 1 | 0 | 0 | 0

26. Secondary Outcome: Change From Baseline in Serum CRP Level Over Time-Double-Blind Induction Phase
Description: Serum samples were collected at indicated time points to measure CRP levels. Baseline value was the latest pre-dose assessment with a non-missing value from Double-Blind Induction study phase. Change from Baseline was calculated as value at specified time point minus Baseline value.
Time Frame: Baseline and Weeks 2, 4, 6, and 10
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Milligrams per liter
Arm/Group | Placebo IV | GSK2831781 450 mg IV | GSK2831781 300 mg IV | GSK2831781 150 mg IV | GSK2831781 45 mg IV
Number analyzed (Participants) | 27 | 48 | 11 | 10 | 8
Milligrams per liter
  Week 2; n=27, 47, 11, 10, 8: number analyzed (Participants) | 27 | 47 | 11 | 10 | 8
  Week 2; n=27, 47, 11, 10, 8 | -1.52 (8.508) | 1.01 (8.004) | 8.23 (16.881) | 25.14 (62.574) | -7.71 (14.627)
  Week 4; n=26,45,7,7,7: number analyzed (Participants) | 26 | 45 | 7 | 7 | 7
  Week 4; n=26,45,7,7,7 | -3.38 (8.188) | 6.73 (21.625) | 0.74 (3.376) | 26.23 (62.003) | -9.41 (18.059)
  Week 6; n=24,45,8,6,8: number analyzed (Participants) | 24 | 45 | 8 | 6 | 8
  Week 6; n=24,45,8,6,8 | -3.09 (6.748) | 4.45 (13.491) | 2.34 (7.016) | 12.20 (15.566) | -8.16 (18.602)
  Week 10; n=22,39,4,4,4: number analyzed (Participants) | 22 | 39 | 4 | 4 | 4
  Week 10; n=22,39,4,4,4 | 2.89 (9.460) | 8.99 (21.549) | 8.40 (8.102) | 6.75 (13.749) | -8.48 (20.407)

27. Secondary Outcome: Ratio to Baseline in Fecal Calprotectin Over Time-Double-Blind Induction Phase
Description: Fecal samples were collected at indicated time points to measure fecal calprotectin. Baseline value was the latest pre-dose assessment with a non-missing value from Double-Blind Induction study phase. Ratio to Baseline is the value at specified time point divided by Baseline value
Time Frame: Baseline and Weeks 2, 4, 6, and 10
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Placebo IV | GSK2831781 450 mg IV | GSK2831781 300 mg IV | GSK2831781 150 mg IV | GSK2831781 45 mg IV
Number analyzed (Participants) | 27 | 48 | 11 | 10 | 8
Ratio
  Week 2; n=25,40,9,9,6: number analyzed (Participants) | 25 | 40 | 9 | 9 | 6
  Week 2; n=25,40,9,9,6 | 1.28 (311.68) | 0.90 (504.70) | 0.57 (206.90) | 2.05 (565.80) | 0.57 (200.43)
  Week 4; n=3,2,0,2,0: number analyzed (Participants) | 3 | 2 | 0 | 2 | 0
  Week 4; n=3,2,0,2,0 | 0.28 (296.27) | 1.58 (794.82) |  | 1.60 (55.72) |
  Week 6; n=23,37,7,6,7: number analyzed (Participants) | 23 | 37 | 7 | 6 | 7
  Week 6; n=23,37,7,6,7 | 0.99 (688.97) | 0.99 (576.84) | 4.01 (8478.60) | 3.42 (477.17) | 2.51 (182.31)
  Week 10; n=20,31,3,3,4: number analyzed (Participants) | 20 | 31 | 3 | 3 | 4
  Week 10; n=20,31,3,3,4 | 1.68 (217.05) | 1.27 (961.25) | 3.82 (76.67) | 8.50 (2110.12) | 0.50 (251.03)

28. Secondary Outcome: Area Under the Concentration-time Curve Over the 1st Dosing Interval (AUC[0-tau]) for GSK2831781 Following SC Dosing in Double-Blind Extended Treatment Phase
Description: Blood samples were collected at indicated time points for pharmacokinetic (PK) analysis of GSK2831781. PK parameters were calculated using standard non-compartmental analysis.
Time Frame: Week 14 (pre-dose, 24, 72 and 168 hours post-dose); Week 18 (pre-dose and early withdrawal post-dose)
Population: Pharmacokinetic Double-Blind Extended Population comprised of all participants in the Safety Extended Treatment Phase population who had at least 1 non-missing PK assessment in the Extended Treatment phase. Only those participants with data at more than two of the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | GSK2831781 300 mg SC
Number analyzed (Participants) | 3
Hours*micrograms per milliliter | 24336.92 (23.797)

29. Secondary Outcome: Maximum Concentration (Cmax) of GSK2831781 Observed Following 1st SC Dosing in Double-Blind Extended Treatment Phase
Description: Blood samples were collected at indicated time points for PK analysis of GSK2831781. PK parameters were calculated using standard non-compartmental analysis.
Time Frame: Week 14 (pre-dose, 24, 72 and 168 hours post-dose); Week 18 (pre-dose and early withdrawal post-dose)
Population: Pharmacokinetic Double-Blind Extended Population. Only those participants with data at more than two of the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | GSK2831781 300 mg SC
Number analyzed (Participants) | 3
Micrograms per milliliter | 55.64 (13.374)

30. Secondary Outcome: Time at Which the Maximum Concentration is Observed (Tmax) for GSK2831781 Following 1st SC Dosing in Double-Blind Extended Treatment Phase
Description: as for outcome 29
Time Frame: Week 14 (pre-dose, 24, 72 and 168 hours post-dose); Week 18 (pre-dose and early withdrawal post-dose)
Population: as for outcome 29
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK2831781 300 mg SC
Number analyzed (Participants) | 3
Hours | 72.03 [24.3 to 170.0]

31. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies at Each Visit-Double-Blind Induction Phase
Description: Serum samples were assessed for the presence of anti-drug antibodies using a tiered approach. The assay involved screening, confirmation and titration steps. If serum samples tested positive in the screening assay, they were considered 'potentially positive' and were further analyzed for the specificity using the confirmation assay. Samples that confirmed positive in the confirmation assay were reported as 'confirmed positive'.
Time Frame: Baseline, Weeks 2, 4, 6, and 10
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo IV | GSK2831781 450 mg IV | GSK2831781 300 mg IV | GSK2831781 150 mg IV | GSK2831781 45 mg IV
Number analyzed (Participants) | 27 | 48 | 11 | 10 | 8
Participants
  Baseline; n=27,48,11,10,8 | 0 | 0 | 0 | 0 | 0
  Week 2; n=27,47,11,10,8: number analyzed (Participants) | 27 | 47 | 11 | 10 | 8
  Week 2; n=27,47,11,10,8 | 0 | 0 | 0 | 0 | 0
  Week 4; n=25,46,7,7,7: number analyzed (Participants) | 25 | 46 | 7 | 7 | 7
  Week 4; n=25,46,7,7,7 | 0 | 0 | 0 | 0 | 0
  Week 6; n=1,3,3,0,3: number analyzed (Participants) | 1 | 3 | 3 | 0 | 3
  Week 6; n=1,3,3,0,3 | 0 | 0 | 0 |  | 0
  Week 10; n=22,39,4,4,4: number analyzed (Participants) | 22 | 39 | 4 | 4 | 4
  Week 10; n=22,39,4,4,4 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Non-SAEs and SAEs were collected up to Week 12 (participants who entered OL induction phase) or Week 14 (participants who entered double-blind ETP) for Double-blind induction phase, from Week 14 to 30 for double-blind ETP, from Week 12 to 22 for OL induction phase and from Week 22 to 42 for OL ETP
Description: Non-SAEs and SAEs were collected in Safety Population for Double-blind induction phase, Safety ETP for double-blind ETP, Safety OL induction and Safety OL ETP for OL induction phase and OL ETP respectively.
Arm/Group | Placebo IV | GSK2831781 450 mg IV | GSK2831781 300 mg IV | GSK2831781 150 mg IV | GSK2831781 45 mg IV | Placebo SC | GSK2831781 300 mg SC | Open-label GSK2831781 450 mg IV | Open-label GSK2831781 300 mg SC
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/48 | 0/11 | 0/10 | 0/8 | 0/5 | 0/8 | 0/42 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/27 | 6/48 | 1/11 | 0/10 | 0/8 | 0/5 | 1/8 | 3/42 | 0/7
Other Adverse Events (participants affected / at risk) | 10/27 | 26/48 | 6/11 | 2/10 | 2/8 | 1/5 | 3/8 | 18/42 | 2/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo IV (N=27) | GSK2831781 450 mg IV (N=48) | GSK2831781 300 mg IV (N=11) | GSK2831781 150 mg IV (N=10) | GSK2831781 45 mg IV (N=8) | Placebo SC (N=5) | GSK2831781 300 mg SC (N=8) | Open-label GSK2831781 450 mg IV (N=42) | Open-label GSK2831781 300 mg SC (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo IV (N=27) | GSK2831781 450 mg IV (N=48) | GSK2831781 300 mg IV (N=11) | GSK2831781 150 mg IV (N=10) | GSK2831781 45 mg IV (N=8) | Placebo SC (N=5) | GSK2831781 300 mg SC (N=8) | Open-label GSK2831781 450 mg IV (N=42) | Open-label GSK2831781 300 mg SC (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 12 (13) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Mixed anxiety and depressive disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somatic symptom disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Myocardial fibrosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malabsorption (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart rate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis toxic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucose urine present (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic venous thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosed varicose vein (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/65/NCT03893565/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/65/NCT03893565/SAP_001.pdf